CLINICAL TRIAL: NCT05606848
Title: Efficacy and Safety of Fresubin Support Drink for Enteral Nutrition Support in Perioperative Patients With Gastrointestinal Cancer: A Prospective, Randomized, Open-Label, Active-Controlled Multi-Center Clinical Trial
Brief Title: To Test the Food for Special Medical Purpose in Perioperative Patients With Gastrointestinal Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fresenius Kabi Sino-Swed Pharmaceutical Corp. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SUPE-001-CEN
Record Dates: First submitted 2022-10-27; First posted 2022-11-07 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Gastrointestinal Cancer
MeSH Terms: conditions — Gastrointestinal Neoplasms | interventions — Food

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control product (Active Comparator): Nutrition Emulsion (TPF-T) is a tumor-specific enteral nutrition therapy
  Interventions: Other: Nutrition Emulsion (TPF-T)
- Study prodcut (Experimental): Foods for special medical purposes [FSMP] for patients with tumors
  Interventions: Other: Foods for special medical purposes [FSMP] for patients with tumors

INTERVENTIONS:
Other: Nutrition Emulsion (TPF-T) — All patients will be randomized to receive the FSMP or control product.
  * Before the surgery: Patients daily intake control product with recommended energy.
  * 1-8 days after surgery: Patients gradually increase control product intake to reach the recommended energy.
  Arms: Control product
Other: Foods for special medical purposes [FSMP] for patients with tumors — All patients will be randomized to receive the FSMP or control product.
  * Before the surgery: Patients daily intake FSMP with recommended energy.
  * 1-8 days after surgery: Patients gradually increase FSMP intake to reach the recommended energy.
  Arms: Study prodcut

SUMMARY:
This is a prospective, randomized, open label, active-controlled, multi-centre, non-inferiority clinical trial. Aim of the study is to evaluate the efficacy and safety of Fresubin Support Drink in patients with gastrointestinal cancer undergoing surgical resection during the perioperative period.

DETAILED DESCRIPTION:
This is a prospective, randomized, open label, active-controlled, multi-centre, non-inferiority clinical trial. The IMP includes study product and control product. The study product will be Fresubin Support Drink (FSMP), the control product will be Enteral Nutrition Emulsion(TPF-T) . Not exceed 350 patients will be randomly assigned to the Fresubin Support Drink (FSMP) group or Enteral Nutrition Emulsion(TPF-T) group at a ratio of 1:1.

Prealbumin, albumin, C-reactive protein (CRP), immunology parameters, vital signs, nutrition and safety-related laboratory parameters, compliance, and Adverse Events (AEs) will be evaluated in this study.

ELIGIBILITY:
Inclusion criteria

1. Agreed to participate in the study with signed ICF;
2. Age 18-75 years;
3. Patient has gastrointestinal cancer confirmed by histological or imagological method and scheduled for resection via open or laparoscopic surgery;
4. Radiotherapy and/or Chemotherapy was not performed within 2 weeks before screening;
5. Hemoglobin ≥ 90 g/L
6. Albumin ≥ 2.5 g/dL
7. BMI ≥18.5 and ≤29 kg/m2;
8. ECOG Performance status 0-2 preoperatively;
9. Expected survival time >6 months.

Exclusion criteria

1. Contraindication or intolerance against EN, e.g., acute gastrointestinal bleeding, ileus (Grade≥3 NCI-CTCAE v 5.0);
2. Any congenital defect of amino acid or carbohydrate metabolism, such as phenylalaninemia, galactosaemia;
3. Conditions requiring emergency surgery;
4. Conditions other than cancer and surgery that can be associated with loss of body weight e.g. serious active clinical infections (> Grade 2, NCI-CTCAE 5.0), including active tuberculosis, or self-reported HIV infection or active hepatitis B or C;
5. Known treatment refractory metabolic disease (e.g., poorly-controlled diabetes mellitus or fasting blood glucose≥ 10mmol/L, hyperthyroidism, hypothyroidism, metabolic acidosis);
6. Cardiac dysfunction (New York Heart Association Functional Class > III);
7. Severe hepatic dysfunction associated with significant increase of AST or ALT > 5 ULN or bilirubin > 3 ULN;
8. Severe renal dysfunction associated with serum creatinine concentration > 1.5 ULN and/or required dialysis;
9. Active treatment refractory bleeding;
10. Other malignancies in the last 3 years (except for successfully treated in situ basocellular skin or in situ cervical uterine tumours);
11. Known disease that could seriously affect the digestion and absorption of the IMPs;
12. History of drug or alcohol abuse within 6 months prior to screening;
13. Current use of medication or nutritional supplements containing more than 500 mg of EPA+DHA/day or fish oil capsules/ supplements containing more than 500 mg EPA + DHA/day at screening;
14. Current use of muscle growth supporting substances (e.g., anabolics) at screening;
15. Planned chemotherapy, radiotherapy or immunotherapy during the first 12 days following the surgical tumor resection;
16. Transfusion of blood products within 1 week before screening;
17. Known allergy to contents of the study product or control product;
18. Pregnancy or lactation;
19. Participation in another clinical study with an investigational drug, FSMP or an investigational medical device one month prior to start of study or planned participation in another clinical trial as specified before during the course of the study period;
20. Patient who is unable to understand the spoken and written information or not willing or not able to comply with scheduled visits and the requirements of the study protocol;
21. Considered not suitable for study participation by the investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2022-11-30 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Change in serum prealbumin | from baseline to close out visit (Post-operation Day 5-8)

SECONDARY OUTCOMES:
Change in body weight (%) | from baseline to Visit 2（Pre-operation Day 1）, Visit 4（Post-operation Day 5 or 6） and close out visit(Post-operation Day 5-8)
Change in serum prealbumin | from baseline to Visit 2（Pre-operation Day 1）, Visit 3（Post-operation Day 1） and Visit 4（Post-operation Day 5 or 6）
Change in serum albumin | from baseline to Visit 3（Post-operation Day 1） and close out visit(Post-operation Day 5-8)
Change in BMI | from baseline to close out visit(Post-operation Day 5-8)
  weight in kilograms, height in meters，weight and height will be combined to report BMI in kg/m^2
Change in PG-SGA | from baseline to Close out Visit(Post-operation Day 5-8)
Change in grip strength | from baseline to Close out Visit(Post-operation Day 5-8)
  hand grip strength measured in kg
Change in CRP | from baseline to Visit 3（Post-operation Day 1） and Close out Visit(Post-operation Day 5-8)
Change in total lymphocyte count | from baseline to Visit 3（Post-operation Day 1） and Close out Visit(Post-operation Day 5-8)
Change in total number of CD4+and CD8+ | from baseline to Visit 3（Post-operation Day 1） and Close out Visit(Post-operation Day 5-8)
Change in CD4+ % and CD8+% | from baseline to Visit 3（Post-operation Day 1） and Close out Visit(Post-operation Day 5-8)
  the respective percentage of CD4+ T lymphocytes and CD8+ T lymphocytes in total lymphocytes
Change in CD4+ T lymphocytes /CD8+ T lymphocytes | from baseline to Visit 3（Post-operation Day 1） and Close out Visit(Post-operation Day 5-8)
Change in neutrophil/lymphocyte ratio | from baseline to Visit 3（Post-operation Day 1） and Close out Visit(Post-operation Day 5-8)
Change in blood glucose | from baseline to Visit 3（Post-operation Day 1） and Close out Visit(Post-operation Day 5-8)
Change in lipids | from baseline to Visit 3（Post-operation Day 1） and Close out Visit(Post-operation Day 5-8)
Change in ECOG performance status | from baseline to Close out Visit(Post-operation Day 5-8)
All adverse events (AEs), including serious adverse events (SAEs) for assessment of safety and tolerability | from baseline to Close out Visit(Post-operation Day 5-8)
Energy intake in kcal / kg BW | from baseline to Close out Visit(Post-operation Day 5-8)
  Total volume of IMP consumed

CONTACTS AND LOCATIONS:
Overall Officials: Hanping Shi, MD, Principal Investigator — Capital Medical University Affiliated Beijing Shijitan Hospital
Locations (14):
- China (14):
  - Beijing Hospital, Beijing
  - Beijing Cancer Hospital, Beijing
  - Capital Medical University Affiliated Beijing Shijitan Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - Xiangya Hospital Central South University, Changsha
  - The First Affiliated Hospital Of Guangzhou Medical University, Guangzhou
  - Nanfang Hospital, Guanzhou
  - Yunnan Cancer Hospital（The affiliated hospital of Kunming medical university）, Kunming
  - Jiangsu Province Hospital of Chinese Medicine, Nanjing
  - The Affiliated Hospital of Qingdao University, Qingdao
  - The Fourth Hospital of Hebei Medical University （Hebei Tumor Hospital）, Shijia Zhuang
  - The First Affiliated Hospital of SOOCHOW University, Suzhou
  - The Central Hospital of Wuhan, Wuhan
  - Union hospital tongji medical college huazhong university of science and technology, Wuhan

IPD SHARING:
Plan to Share IPD: No